CLINICAL TRIAL: NCT03107715
Title: Assessing the Feasibility of a Breastfeeding Champion Intervention and a Positive Messaging Module During the Prenatal Period - a Pilot
Brief Title: Prenatal Interventions to Promote Exclusive Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lydia Furman (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Mt. Sinai Health Care Foundation (Other)
Responsible Party: Sponsor-Investigator, Lydia Furman, Professor of Pediatrics, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 04-17-04
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Breastfeeding; Intention; Health Behavior
Keywords: exclusive breastfeeding; health disparity; prenatal intervention
MeSH Terms: conditions — Breast Feeding; Health Behavior

STUDY DESIGN:
Intervention Model Description: Sequential presentation of 2 prototype interventions with pre/post test and follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Champion (Active Comparator): The Breastfeeding Champion Intervention (Intervention A) utilizes information about Breastfeeding Champions from the Coffective™ program: participants will be guided to tap and scroll through the content and will receive a follow up handout and encouragement to select a Champion.
  Interventions: Behavioral: Breastfeeding Champion
- Positive Messaging (Active Comparator): The Positive Messaging Intervention (Intervention B) utilizes positive messaging from several sources and is modelled on the WIC Loving Support™ approach: participants will click on (istock-purchased) photographs which each reveal an informational statement about exclusive breastfeeding benefits and tips, followed by receipt of a summary handout.
  Interventions: Behavioral: Positive Messaging

INTERVENTIONS:
Behavioral: Breastfeeding Champion — iPad-based behavioral intervention facilitated by researcher
  Arms: Breastfeeding Champion
Behavioral: Positive Messaging — iPad based behavioral intervention facilitated by researcher
  Arms: Positive Messaging

SUMMARY:
Background: Exclusive breastfeeding through age 6 months is the optimal infant feeding method due to lifesaving benefits for children and mothers (AAP, others). Exclusive breastfeeding in-hospital is critical because in-hospital formula supplementation doubles risk of non-exclusive breastfeeding at 30-60 days (Chantry et al, 2014). While breastfeeding initiation rates have increased at our inner-city Baby Friendly - designated maternity hospital, exclusive breastfeeding lags. CDC mPINC data (maternity practices in infant nutrition and care, 2015) demonstrate this is a national problem, with >50% of surveyed hospitals endorsing supplementation of "10-49%" of breastfed infants.

Study Objective: The study objective is to evaluate acceptance/satisfaction of 2 prenatal interventions (breastfeeding champion and positive messaging) and to determine if these affect exclusive breastfeeding intention and practice.

Methods: In this prospective intervention study with follow-up chart review, we will pilot two 5-minute-long iPad-based interventions for 1 month each in obstetrical clinics, following a required 28-week obstetrical visit breastfeeding education. All expectant mothers (including 14-17 year olds with guardian) are eligible. Outcomes are acceptance (enrollment rate), satisfaction (Likert-based), impact on exclusive breastfeeding intention (pre/post query) and secondarily impact on exclusive breastfeeding in-hospital and at 2 weeks.

DETAILED DESCRIPTION:
Relevance:

This research is aligned with efforts to decrease infant mortality and associated racial disparities via culturally competent interventions, and our aim is that it will be possible to model a larger intervention trial using the data generated in this pilot study. The project showcases work which is clinically meaningful, addresses an important racial health disparity in a vulnerable population (predominantly African-American expectant women) and is allied with hospital quality measures (PC-05, exclusive breastfeeding in hospital).

Background:

Exclusive breastfeeding through age 6 months is the optimal infant feeding method due to lifesaving benefits for children and mothers (AAP, others). Exclusive breastfeeding in-hospital is critical because in-hospital formula supplementation doubles risk of non-exclusive breastfeeding at 30-60 days (Chantry et al, 2014). While breastfeeding initiation rates have increased at our inner-city Baby Friendly - designated maternity hospital, exclusive breastfeeding lags. CDC mPINC data (maternity practices in infant nutrition and care, 2015) demonstrate this is a national problem, with >50% of surveyed hospitals endorsing supplementation of "10-49%" of breastfed infants.

Study Objective and Aims:

The study objective is to evaluate acceptance/satisfaction of 2 prenatal interventions (breastfeeding champion and positive messaging) and to determine if these affect exclusive breastfeeding intention and practice.

Study Aims are "1." To determine if intention to exclusively breastfeed changes from before to after the intervention is implemented "2." To determine the acceptance and satisfaction of the interventions "3." To determine and compare the rates of exclusive breastfeeding in-hospital and at 2-weeks postpartum among women who received the champion and positive messaging interventions

Methods:

Study Design: The study is a pretest-posttest sequential group design chosen to evaluate the effect of two prenatal breastfeeding interventions on exclusive breastfeeding intention. Intervention A (Breastfeeding Champion) and Intervention B (Positive Messaging) will be administered during months 1 and 2, respectively, of the study.

Population and Setting: The setting is University Hospitals MacDonald Women's Hospital, an academic tertiary care birthing center in urban Cleveland, OH with approximately 3,800 deliveries per year. The eligible population includes expectant women ages 14 years and up (with guardian present if ages 14-17 years) who are attending a prenatal visit at an on-site clinic and have completed required breastfeeding education presented at or before 28 weeks of gestation. The clinics serve a predominantly African-American WIC-eligible population.

Interventions: Both interventions use a secured and protected iPad, and the total interaction with the participant will take about 10 minutes. Intervention A utilizes information about Breastfeeding Champions from the Coffective™ program: participants will be guided to tap and scroll through the content and will receive a follow up handout and encouragement to select a Champion. Intervention B utilizes positive messaging from several sources and is modelled on the WIC Loving Support™ approach: participants will click on (istock-purchased) photographs which each reveal an informational statement about exclusive breastfeeding benefits and tips, followed by receipt of a summary handout.

Data Collection: After informed consent is obtained, sociodemographic information and a pretest to include feeding intention will be administered. Then following the 5-8 minute iPad-based intervention, a short posttest will be administered, which asks a Likert based question about intervention satisfaction and about feeding intention post-intervention. Postpartum, actual feeding method in hospital and at 2 weeks will be gathered by chart review. REDCap will be utilized for data entry.

Outcome Measures: These will reflect the aims:

"1." Intention to exclusively breastfeed post-intervention "2." Likert-based satisfaction with intervention received "3." Rates of exclusive breastfeeding in-hospital and at 2 weeks post-partum

Data Collection Tools: These were created by the study team.

Data analysis and Sample Size considerations:

Sample size - Aim #1 of the study is to determine if intention to exclusively breastfeed changes from before to after the interventions are implemented. There are no published data on this question utilizing these interventions with which to formulate a hypothesis and perform the requisite sample size to test that hypothesis. This will be considered a hypothesis generating study and feasibility of enrollment will determine the sample size. We will approach all eligible women during 2-month study period. We anticipate that approximately 31 women per week will be eligible, of whom approximately 80% will agree to participate, and over a 2-month study period, 250 women could be enrolled.

Data analysis - Nominal variables will be described using frequencies and percentages. Normally distributed continuous variables will be described using means and standard deviations, and non-normally distributed continuous variables will be described using medians and IQRs (interquartile ranges). We will compare nominal variables, e.g. those who received differing interventions (champion versus positive messaging) using Chi squared analyses or Fisher's exact test as appropriate. Distributionally appropriate two-sample tests will be used to compare continuous variables. Additional analyses may be carried out as the data indicate, and will be considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Expectant women receiving prenatal care at UH MacDonald Women's Health Clinic or MAC1200 CLinic
* Completed required breastfeeding education presented at or before 28 weeks of gestation
* Age 14 - 17 years must have guardian/parent present who consents to teen participation, and teen must then assent to participation
* Ages 18 years and older must consent to participate

Exclusion Criteria:

* Medical indication for use of formula only after delivery including HIV+ or will require chemotherapy treatment

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — must be an expectant woman - self-representation of gender identity is required
Enrollment: 243 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Farr, BSE, Principal Investigator — CWRU SOM
Locations (1):
- University Hospital MacDonald Women's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breastfeeding Champion | Positive Messaging
Started | 132 | 111
Completed | 128 | 104
Not Completed | 4 | 7
Not completed — did not deliver at the home hospital | 4 | 6
Not completed — infant stillborn | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breastfeeding Champion | Positive Messaging | Total
Number analyzed (Participants) | 132 | 111 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 129 | 110 | 239
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (4.3) | 24.4 (4.4) | 24.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 111 | 243
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 127 | 99 | 226
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 132 | 111 | 243
marital status [Count of Participants; unit: Participants] — Measure is the number of participants who stated they are married.
  Participants | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Intended to Exclusively Breastfeed Post-intervention
Description: Single query "How do you plan to feed your baby?" with 4 possible responses Just formula / Both breastmilk and formula / Just breastmilk / Unsure
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Breastfeeding Champion | Positive Messaging
Number analyzed (Participants) | 132 | 111
Participants
  Number who intended to exclusively breastfeed | 40 | 36
  Did not intend to exclusively breastfeed | 86 | 67
  Missing information | 2 | 1
  Did not deliver at home hospital | 4 | 6
  stillbirth | 0 | 1

2. Primary Outcome: Number of Participants Who Reported Their Intervention as "Very Interesting" (Response=5) on a 5 Point Likert Scale
Description: Single 5 point Likert scale with query "Was the intervention you received interesting and enjoyable?" Analyzed as all those who said 5 "very interesting" on a 5 point Likert scale; higher score indicates the participant liked/was more interested in the intervention; minimum score =1, maximum score = 5; No scale title - Question was: Was the intervention you received interesting and enjoyable? Please give us your overall impression on a scale from 1-5!
Time Frame: 15 minutes
Measure: Number; unit: participants
Arm/Group | Breastfeeding Champion | Positive Messaging
Number analyzed (Participants) | 132 | 111
participants | 89 | 58

3. Secondary Outcome: Number of Participants Who Exclusively Breastfed In-hospital
Description: Was infant fed breastmilk only in-hospital postpartum (yes/no)
Time Frame: 2 days
Population: Only able to include those who delivered at the home hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Breastfeeding Champion | Positive Messaging
Number analyzed (Participants) | 128 | 104
Participants | 79 | 66

4. Secondary Outcome: Number of Participants Who Exclusively Breastfed at 2 Weeks Postpartum
Description: Was infant fed breastmilk only at 2 weeks postpartum (yes/no)
Time Frame: 2 weeks
Population: those with feeding data at 2 weeks, 68 total missing for Champion and 46 total missing for Positive Messaging
Measure: Count of Participants; unit: Participants
Arm/Group | Breastfeeding Champion | Positive Messaging
Number analyzed (Participants) | 64 | 65
Participants | 26 | 29

ADVERSE EVENTS:
Time Frame: 24 months
Description: no study related adverse events;
Arm/Group | Breastfeeding Champion | Positive Messaging
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/111
Serious Adverse Events (participants affected / at risk) | 0/132 | 1/111
Other Adverse Events (participants affected / at risk) | 0/132 | 0/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breastfeeding Champion (N=132) | Positive Messaging (N=111)
still birth (Pregnancy, puerperium and perinatal conditions) | 0 | 1

LIMITATIONS AND CAVEATS:
This was not a randomized controlled trial - there were no control subjects - this was an active comparator trial and participants were enrolled in non-random blocks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03107715/Prot_SAP_000.pdf